CLINICAL TRIAL: NCT07011446
Title: Usability Evaluation of the Safer Seat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Faieta (Other)
Responsible Party: Sponsor-Investigator, Julie Faieta, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY24090134
Record Dates: First submitted 2025-05-20; First posted 2025-06-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-05

CONDITIONS: Impaired Mobility; Impaired Balance
Keywords: Transfers; Mobility Aid; Mobility Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Safer Seat Trial (Experimental): This study utilizes a single arm design per the goals of the usability trial. The intervention centers on trialing vehicle seat transfers with and without the Safer Seat.
  Interventions: Device: Safer Seat Usability Trial

INTERVENTIONS:
Device: Safer Seat Usability Trial — Participants will be asked to transfer onto/off of the vehicle seat using their normal method of transfer and then to trial transferring onto/off of a vehicle seat with the Safer Seat 1 one or more times with study personnel. Demographic data will be recorded for all participants to include age, sex, and type of mobility disability. Transfers will be observed by the research personnel and success in transfers will be recorded according to the Physical Mobility Scale.
  Usefulness and usability of the Safer Seat transfer experience will be reported by participants via Technology Acceptance Model Surveys; and participants will engage in a brief semi structured interview that will be audio recorded and transcribed via Microsoft Teams.

SUMMARY:
This is an initial usability assessment of a vehicle Seat Transfer device, the Safer Seat. The study will involve target end users (individuals with mobility impairments) trialing the Safer Seat and providing feedback via the Technology Acceptance Model Survey's Modified from Davis (1985) and brief qualitative interview.

DETAILED DESCRIPTION:
This study investigates the initial usability of the Safer Seat vehicle transfer aid. Participants with impaired mobility, strength, or balance are being asked to transfer onto and off of a vehicle seat with and without the device to trial its usability. In addition, transfers are doing rated by a licensed occupational therapist according to the Physical Mobility Scale to determine if independence level is affected. Usability evaluation is being done both qualitatively and quantitatively using Technology Assessment Surveys and a semi-structured interview. Insight gained through this initial trial will be used to refine the design of the Safer Seat.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Currently living with impaired mobility, strength, or balance
* Self-reported ability to complete transfers at modified independent (independent with the use of an assistive device) or minimal assist (a small amount of assistance from another person) level

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Physical Mobility Scale | Day 1
  Used to rate ability level in sit to stand and stand to sit transfers from 0 if not able to bear weight, to 5 if independent and not needing to use upper extremities for assistance.

SECONDARY OUTCOMES:
Technology Acceptance Model Perceived Ease of Use, Usefulness, and Attitudes Toward Use questionnaires | Day 1
  Modified from Davis (1985) surveys to assess Perceived Ease of Use, Perceived Usability, and Attitudes Toward. Survey item responses on 5-item likert scale. Scoring progresses from Strongly Disagree (1) to Strongly Agree (5). For most items "Strongly Agree" indicase the individual favors the intervention. There are a few items phrased in a negative manner such that a response of "Strongly Disagree" indicates the individual favors the intervention; these items are reverse coded when scoring.
Semi structured interview | Day 1
  Questions were focused on the usability and usefulness of the Safer Seat.
Demographic Data | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Julie Faieta, PhD, MOT, Principal Investigator — University of Pittsburgh
Locations (1):
- Univeristy of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No